CLINICAL TRIAL: NCT07086105
Title: A Phase 1, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Preliminary Efficacy of Intratumoural Adze1.C in Participants With Metastatic Melanoma
Brief Title: A Study to Evaluate Adze1.C in Participants With Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adze Biotechnology Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Adze Biotechnology Inc (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADZE1.C-001
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adze1.C Dose Escalation (Experimental): Participants will receive Adze1.C by intratumoural injection. All will begin with a low seroconversion dose (1 million viral particles), followed three weeks later by an escalation dose based on cohort assignment:
  Cohort 1: 100 million vp Cohort 2: 1 billion vp Cohort 3: 10 billion vp Doses are given every two weeks for up to 14 weeks. Dose escalation follows a 3+3 design to evaluate safety, tolerability, and early signs of efficacy.
  Interventions: Drug: Adze1.C

INTERVENTIONS:
Drug: Adze1.C — Conditionally replicative oncolytic adenovirus expressing CD40L, administered by intratumoural injection in dose escalation cohorts.

SUMMARY:
This is Phase I, open label, multi-center clinical trial evaluating an investigational treatment, Adze1.C. Adze1.C is a type of oncolytic virus therapy for adults with advanced Melanoma that have not responded to standard treatments. Oncolytic viruses are designed to infect and destroy cancer cells and have the potential to stimulate the immune system to fight tumors. The purpose of this study is to determine the safety of Adze1.C, how well it is tolerated, and to identify the highest dose that can be safely given.

DETAILED DESCRIPTION:
This Phase 1, multicenter, open-label, dose-escalation study is designed to evaluate the safety, tolerability, pharmacodynamics, and preliminary efficacy of Adze1.C, a conditionally replicative oncolytic adenovirus encoding CD40L, in participants with metastatic melanoma.

Up to 30 participants will be enrolled across three sequential dose cohorts. All participants will first receive a low initial (seroconversion) dose of Adze1.C injected directly into their tumour. Three weeks later, they will receive a higher dose based on their assigned cohort:

cohort 1: Adze1.C 1 × 10E8 vp

cohort 2: Adze1.C 1 × 10E9 vp

cohort 3: Adze1.C 1 × 10E10 vp

Dose escalation will follow a standard 3+3 design. Participants will be closely monitored for side effects for five weeks after the first injection. Those who tolerate the treatment may receive additional doses every two weeks for up to 14 weeks total.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older at Screening.
2. Histologically confirmed unresectable Stage IIIB to IV metastatic melanoma.
3. Refractory to, or unsuitable for, standard treatment options as determined by the investigator.
4. Not a suitable candidate for curative resection.
5. Presence of measurable disease per iRECIST (excluding irradiated lesions unless progression post-radiation is documented).
6. ECOG performance status of 0 or 1 at Screening.
7. Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Uncontrolled intercurrent illness, including but not limited to:

   * Active systemic infection or fever ≥ 38°C within 5 days prior to Screening
   * Symptomatic congestive heart failure
   * NYHA Class III or IV heart failure
   * Unstable angina or arrhythmia
   * Psychiatric illness or social conditions that limit compliance
2. Immunocompromised status or known HIV infection with ongoing antiretroviral therapy.
3. Active or clinically significant liver disease, including:

   * Hepatitis B surface antigen (HBsAg) positive
   * Hepatitis C virus RNA positive
4. History of organ transplantation.
5. Prior treatment with adenovirus therapy.
6. Prior oncolytic virus treatment within 2 months of Screening.
7. Use of systemic immunosuppressants or immune-modifying drugs at Screening or planned during study.
8. Use of cidofovir within 14 days of Adze1.C dosing.
9. Any other condition which, in the investigator's judgment, would make the participant inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | From Day 1 (first dose) through Week 16 (end of treatment visit)
  Safety will be assessed based on the frequency, nature, and severity of TEAEs, graded per CTCAE v5.0.
Incidence of dose-limiting toxicities (DLTs) | Week 1 Day 1 to Week 6 Day 1 (5-week DLT evaluation period)
  Number of participants who experience DLTs during the 5-week period following the seroconversion and escalation doses, per predefined DLT criteria.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) determination | Through Week 16
  RP2D will be determined by the Safety Review Committee (SRC) based on cumulative safety, DLT, and tolerability data from all cohorts.
Detection of viral shedding in bodily fluids | From Day 1 through Week 16
  Presence of Adze1.C viral particles will be assessed in serum, saliva, stool, and urine using PCR-based methods.
Objective response rate (ORR) | From first dose through disease progression (estimated up to 6 months)
  Proportion of participants with complete or partial response, assessed per iRECIST.
Progression-Free Survival (PFS) | From first dose to disease progression or death (estimated up to 12 months)
  Time from first treatment to documented disease progression or death from any cause, per iRECIST.
Patient-reported quality of life using EORTC QLQ-C30 | From baseline to Week 16
  The EORTC QLQ-C30 is a widely used and validated 30-item questionnaire used to assess quality of life (QoL) in cancer patients. Scores are transformed to a 0-100 scale. For functional scales and global health status/QoL, higher scores indicate better functioning or quality of life. For symptom scales/items, higher scores reflect greater symptom burden (i.e., worse outcome).

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Tasman Oncology Research, Southport, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No